CLINICAL TRIAL: NCT01981941
Title: Post-marketing Clinical Study of Gabapentin Enacarbil -Non-blinded Study in Restless Legs Syndrome (RLS) Patients With Moderate Renal Impairment-
Brief Title: Post-marketing Study of Gabapentin Enacarbil to Evaluate the Effect in Restless Leg Syndrome (RLS) Patients With Moderate Renal Impairment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8825-CL-0103
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Restless Legs Syndrome (RLS)
Keywords: Gabapentin; Restless legs syndrome (RLS)
MeSH Terms: conditions — Restless Legs Syndrome | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): Oral
  Interventions: Drug: Gabapentin enacarbil

INTERVENTIONS:
Drug: Gabapentin enacarbil — Oral

SUMMARY:
To evaluate the safety, efficacy and pharmacokinetics of gabapentin enacarbil in moderate to severe primary RLS patients with moderate renal impairment and to confirm dosage and administration in such population.

DETAILED DESCRIPTION:
This study is a multicenter, non-blinded, non-comparative study. Patients who meet the eligible criteria will undergo one week observation period followed by four week treatment period. In treatment period, patients will receive gabapentin enacarbil orally one daily after dinner. After the four-week treatment period with gabapentin enacarbil, a one-week post-observation period will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with restless legs syndrome (RLS) according to the international RLS Study Group Diagnostic Criteria
* Patients whose score is 15 or greater on the International RLS (IRLS) Rating Scale on the first day of the pre-observation period.
* Patients whose creatinine clearance level at the first day of pre-observation period is ≥30 mL/min to <60mL/min estimated by Cockcroft-Gaul t equation
* Patients who provide written consent

Exclusion Criteria:

* Patients with sleep disorder such as sleep apnea syndrome, which affects the RLS evaluation
* Patients with history of augmentation and treatment rebound of RLS symptoms when using dopamine agonis
* Patients with neuropathy and movement disorder (diabetic neuropathy, Parkinson's disease, multiple sclerosis, dyskinesia, rheumatoid arthritis etc)
* Patients with uncontrolled diabetes [HbA1c>7.5% (NGSP value), in the past six months], iron deficiency anemia, or drug administration of hypnotic sedatives.
* Patients who attempted suicide within six months prior to the consent obtained, or who have been diagnosed as a suicide risk by investigator or sub-investigator
* Patients with moderate or severe depression
* Patients with alcohol dependence or drug intoxication or who have a history of abuse or drug dependence in the past one year
* Patients whose job is shift work, professional driver, or engaging in hazardous activities such as operating machinery
* Patients with history of hypersensitivity to gabapentin
* Patients who have experience to participate in other post-marketing clinical studies or clinical trials within 12 weeks prior to the start of pre-observation
* Others: patients who are concluded to be ineligible by an investigator or sub-investigator as ineligible

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2015-05-13 (Actual); Study Completion 2015-05-13 (Actual)

PRIMARY OUTCOMES:
Change in International Restless Leg Syndrome (IRLS) rating scale score | Baseline and at 4 week of the treatment (or at discontinuation)

SECONDARY OUTCOMES:
Change in Investigator-rated clinical global impression (ICGI) score | Baseline and at 4 week of the treatment (or at discontinuation)
Change in Patient-related clinical global impression (PCGI) score | Baseline and at 4 week of the treatment (or at discontinuation)
  Baseline and at 4 week of the treatment (or at discontinuation)
Safety assessed by the incidence of adverse events, vital signs, labo-tests, body weight and Epworth sleepiness scale | Up to 5 weeks
Plasma gabapentin concentration | Up to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Principal Investigator — Astellas Pharma Inc
Locations (5):
- Japan (5):
  - Chugoku
  - Chūbu
  - Kansai
  - Kanto
  - Kyushu

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=147